CLINICAL TRIAL: NCT05687578
Title: A Prospective, Non-Randomized, Multi-Center Observational Study to Establish a Physical Baseline Profile for Individual Study Subjects Using Various Modalities and Identify Deviations Via Longitudinal Monitoring That May Develop Over Time
Brief Title: PUER ("Previously Unrecognized Emerging Risks") Life Clinical Study
Acronym: PUER
Status: Enrolling by invitation | Type: Observational
Sponsor: Puer Research, LLC (Network)
Responsible Party: Sponsor
Other Study IDs: PLI001
Record Dates: First submitted 2023-01-03; First posted 2023-01-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Aging
Keywords: Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, including genomic samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurements Only — This is an observational study only using biospecimen and imaging-based measurements only

SUMMARY:
This is a minimal risk, prospective, non-randomized, multi-center population based observational study to establish a physical baseline profile for individual study subjects using various modalities (blood draws, non-invasive imaging, stool samples, saliva samples) and identify deviations through longitudinal monitoring that may develop over time and may be relevant to human health and healthy longevity.

DETAILED DESCRIPTION:
The two key elements of the PUER Research protocol include (1) molecular and laboratory profiling and (2) non-invasive imaging and wearables/ "quantified self" measurements. All elements are optional. Molecular assessments will be conducted using peripheral blood samples, and potentially urine, stool or saliva samples. Non-invasive imaging assessment will consist of magnetic resonance imaging (MRI) and computerized tomography (CT) scans, ultrasound, and x-ray. All imaging modalities are optional. Other functional assessments, including respiratory, cardiac and other functions, as well as self-quantifiable assessments via wearables, may also be conducted and are optional.

The study will result in longitudinal data collection to inform if any modalities employed here can inform of baseline deviations for individuals. Researchers at study sites will not be blinded to the data being collected during this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female; age 18 to 90
* Absence or presence of any medical history or any signs or symptoms of any disease
* Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at all visits

Exclusion Criteria:

* Unwillingness or inability to participate in the study
* Unwillingness or inability to provide written Informed Consent Form
* WOCBP with positive pregnancy test at enrollment or at any visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective, population-based observational study. Participants may be recruited from clinical sites that are actively participating in the PUER Research comprehensive evaluation model. Participants and all participating health care providers are unblinded.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Biomarkers that exhibit significant change | 12 Months
  The number of biomarkers that exhibit significant change from baseline to any follow-up timepoint, if obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Szilard Voros, MD, Principal Investigator — Puer Life
Locations (1):
- Puer Research, LLC, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amendola LM, Dorschner MO, Robertson PD, Salama JS, Hart R, Shirts BH, Murray ML, Tokita MJ, Gallego CJ, Kim DS, Bennett JT, Crosslin DR, Ranchalis J, Jones KL, Rosenthal EA, Jarvik ER, Itsara A, Turner EH, Herman DS, Schleit J, Burt A, Jamal SM, Abrudan JL, Johnson AD, Conlin LK, Dulik MC, Santani A, Metterville DR, Kelly M, Foreman AK, Lee K, Taylor KD, Guo X, Crooks K, Kiedrowski LA, Raffel LJ, Gordon O, Machini K, Desnick RJ, Biesecker LG, Lubitz SA, Mulchandani S, Cooper GM, Joffe S, Richards CS, Yang Y, Rotter JI, Rich SS, O'Donnell CJ, Berg JS, Spinner NB, Evans JP, Fullerton SM, Leppig KA, Bennett RL, Bird T, Sybert VP, Grady WM, Tabor HK, Kim JH, Bamshad MJ, Wilfond B, Motulsky AG, Scott CR, Pritchard CC, Walsh TD, Burke W, Raskind WH, Byers P, Hisama FM, Rehm H, Nickerson DA, Jarvik GP. Actionable exomic incidental findings in 6503 participants: challenges of variant classification. Genome Res. 2015 Mar;25(3):305-15. doi: 10.1101/gr.183483.114. Epub 2015 Jan 30. PMID 25637381
- [Background] Arnoldi E, Gebregziabher M, Schoepf UJ, Goldenberg R, Ramos-Duran L, Zwerner PL, Nikolaou K, Reiser MF, Costello P, Thilo C. Automated computer-aided stenosis detection at coronary CT angiography: initial experience. Eur Radiol. 2010 May;20(5):1160-7. doi: 10.1007/s00330-009-1644-7. Epub 2009 Nov 5. PMID 19890640
- [Background] Assarsson E, Lundberg M, Holmquist G, Bjorkesten J, Thorsen SB, Ekman D, Eriksson A, Rennel Dickens E, Ohlsson S, Edfeldt G, Andersson AC, Lindstedt P, Stenvang J, Gullberg M, Fredriksson S. Homogenous 96-plex PEA immunoassay exhibiting high sensitivity, specificity, and excellent scalability. PLoS One. 2014 Apr 22;9(4):e95192. doi: 10.1371/journal.pone.0095192. eCollection 2014. PMID 24755770
- [Background] Bennuru S, Lustigman S, Abraham D, Nutman TB. Metabolite profiling of infection-associated metabolic markers of onchocerciasis. Mol Biochem Parasitol. 2017 Jul;215:58-69. doi: 10.1016/j.molbiopara.2017.01.008. Epub 2017 Feb 8. PMID 28188804
- [Background] Bromberg Y. Building a genome analysis pipeline to predict disease risk and prevent disease. J Mol Biol. 2013 Nov 1;425(21):3993-4005. doi: 10.1016/j.jmb.2013.07.038. Epub 2013 Aug 5. PMID 23928561
- [Background] Chong CA, Tomlinson G, Chodirker L, Figdor N, Uster M, Naglie G, Krahn MD. An unadjusted NNT was a moderately good predictor of health benefit. J Clin Epidemiol. 2006 Mar;59(3):224-33. doi: 10.1016/j.jclinepi.2005.08.005. PMID 16488352
- [Background] Crick F. Central dogma of molecular biology. Nature. 1970 Aug 8;227(5258):561-3. doi: 10.1038/227561a0. No abstract available. PMID 4913914
- [Background] David CEB, Lucas AMB, Cunha PLO, Viana YIP, Yoshinaga MY, Miyamoto S, Filho ABC, Varela ALN, Kowaltowski AJ, Facundo HT. Calorie restriction changes lipidomic profiles and maintains mitochondrial function and redox balance during isoproterenol-induced cardiac hypertrophy. J Physiol Biochem. 2022 Feb;78(1):283-294. doi: 10.1007/s13105-021-00863-4. Epub 2022 Jan 13. PMID 35023023
- [Background] Design and baseline results of the Scandinavian Simvastatin Survival Study of patients with stable angina and/or previous myocardial infarction. Am J Cardiol. 1993 Feb 15;71(5):393-400. doi: 10.1016/0002-9149(93)90438-i. PMID 8430625
- [Background] Dorschner MO, Amendola LM, Turner EH, Robertson PD, Shirts BH, Gallego CJ, Bennett RL, Jones KL, Tokita MJ, Bennett JT, Kim JH, Rosenthal EA, Kim DS; National Heart, Lung, and Blood Institute Grand Opportunity Exome Sequencing Project; Tabor HK, Bamshad MJ, Motulsky AG, Scott CR, Pritchard CC, Walsh T, Burke W, Raskind WH, Byers P, Hisama FM, Nickerson DA, Jarvik GP. Actionable, pathogenic incidental findings in 1,000 participants' exomes. Am J Hum Genet. 2013 Oct 3;93(4):631-40. doi: 10.1016/j.ajhg.2013.08.006. Epub 2013 Sep 19. PMID 24055113
- [Background] Fest J, Vijfhuizen LS, Goeman JJ, Veth O, Joensuu A, Perola M, Mannisto S, Ness-Jensen E, Hveem K, Haller T, Tonisson N, Mikkel K, Metspalu A, van Duijn CM, Ikram A, Stricker BH, Ruiter R, van Eijck CHJ, van Ommen GB, 't Hoen PAC. Search for Early Pancreatic Cancer Blood Biomarkers in Five European Prospective Population Biobanks Using Metabolomics. Endocrinology. 2019 Jul 1;160(7):1731-1742. doi: 10.1210/en.2019-00165. PMID 31125048
- [Background] Ganz P, Heidecker B, Hveem K, Jonasson C, Kato S, Segal MR, Sterling DG, Williams SA. Development and Validation of a Protein-Based Risk Score for Cardiovascular Outcomes Among Patients With Stable Coronary Heart Disease. JAMA. 2016 Jun 21;315(23):2532-41. doi: 10.1001/jama.2016.5951. PMID 27327800
- [Background] Gold L, Ayers D, Bertino J, Bock C, Bock A, Brody EN, Carter J, Dalby AB, Eaton BE, Fitzwater T, Flather D, Forbes A, Foreman T, Fowler C, Gawande B, Goss M, Gunn M, Gupta S, Halladay D, Heil J, Heilig J, Hicke B, Husar G, Janjic N, Jarvis T, Jennings S, Katilius E, Keeney TR, Kim N, Koch TH, Kraemer S, Kroiss L, Le N, Levine D, Lindsey W, Lollo B, Mayfield W, Mehan M, Mehler R, Nelson SK, Nelson M, Nieuwlandt D, Nikrad M, Ochsner U, Ostroff RM, Otis M, Parker T, Pietrasiewicz S, Resnicow DI, Rohloff J, Sanders G, Sattin S, Schneider D, Singer B, Stanton M, Sterkel A, Stewart A, Stratford S, Vaught JD, Vrkljan M, Walker JJ, Watrobka M, Waugh S, Weiss A, Wilcox SK, Wolfson A, Wolk SK, Zhang C, Zichi D. Aptamer-based multiplexed proteomic technology for biomarker discovery. PLoS One. 2010 Dec 7;5(12):e15004. doi: 10.1371/journal.pone.0015004. PMID 21165148
- [Background] Guttmacher AE, Collins FS. Welcome to the genomic era. N Engl J Med. 2003 Sep 4;349(10):996-8. doi: 10.1056/NEJMe038132. No abstract available. PMID 12954750
- [Background] Han X, Aslanian A, Yates JR 3rd. Mass spectrometry for proteomics. Curr Opin Chem Biol. 2008 Oct;12(5):483-90. doi: 10.1016/j.cbpa.2008.07.024. PMID 18718552
- [Background] Hayden EC. Technology: The $1,000 genome. Nature. 2014 Mar 20;507(7492):294-5. doi: 10.1038/507294a. No abstract available. PMID 24646979
- [Background] Lemaitre G, Marti R, Freixenet J, Vilanova JC, Walker PM, Meriaudeau F. Computer-Aided Detection and diagnosis for prostate cancer based on mono and multi-parametric MRI: a review. Comput Biol Med. 2015 May;60:8-31. doi: 10.1016/j.compbiomed.2015.02.009. Epub 2015 Feb 20. PMID 25747341
- [Background] Li J, Huang A, Yao J, Liu J, Van Uitert RL, Petrick N, Summers RM. Optimizing computer-aided colonic polyp detection for CT colonography by evolving the Pareto fronta. Med Phys. 2009 Jan;36(1):201-12. doi: 10.1118/1.3040177. PMID 19235388
- [Background] Netto, G., & Kaul, K, e. (2019). Genomic Applications in Pathology. Springer International Publishing
- [Background] Onal S, Lai-Yuen S, Bao P, Weitzenfeld A, Hart S. Fully automated localization of multiple pelvic bone structures on MRI. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:3353-6. doi: 10.1109/EMBC.2014.6944341. PMID 25570709
- [Background] Randomised trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S). Lancet. 1994 Nov 19;344(8934):1383-9. PMID 7968073
- [Background] Rosenberg S, Elashoff MR, Beineke P, Daniels SE, Wingrove JA, Tingley WG, Sager PT, Sehnert AJ, Yau M, Kraus WE, Newby LK, Schwartz RS, Voros S, Ellis SG, Tahirkheli N, Waksman R, McPherson J, Lansky A, Winn ME, Schork NJ, Topol EJ; PREDICT (Personalized Risk Evaluation and Diagnosis in the Coronary Tree) Investigators. Multicenter validation of the diagnostic accuracy of a blood-based gene expression test for assessing obstructive coronary artery disease in nondiabetic patients. Ann Intern Med. 2010 Oct 5;153(7):425-34. doi: 10.7326/0003-4819-153-7-201010050-00005. PMID 20921541
- [Background] Scaria V. Personal genomes to precision medicine. Mol Cytogenet. 2014 Jan 21;7(Suppl 1 Proceedings of the International Conference on Human):I28. doi: 10.1186/1755-8166-7-S1-I28. eCollection 2014. No abstract available. PMID 24949091
- [Background] Schork NJ. Personalized medicine: Time for one-person trials. Nature. 2015 Apr 30;520(7549):609-11. doi: 10.1038/520609a. No abstract available. PMID 25925459
- [Background] Uppot, R.N., Boas, G., & Flores, E. (2018). Current Developments in Artificial Intelligence and Diagnostic Imaging
- [Background] Yang Q, Li L, Zhang J, Shao G, Zhang C, Zheng B. Computer-aided diagnosis of breast DCE-MRI images using bilateral asymmetry of contrast enhancement between two breasts. J Digit Imaging. 2014 Feb;27(1):152-60. doi: 10.1007/s10278-013-9617-4. PMID 24043592
- [Background] Yet I, Menni C, Shin SY, Mangino M, Soranzo N, Adamski J, Suhre K, Spector TD, Kastenmuller G, Bell JT. Genetic Influences on Metabolite Levels: A Comparison across Metabolomic Platforms. PLoS One. 2016 Apr 13;11(4):e0153672. doi: 10.1371/journal.pone.0153672. eCollection 2016. PMID 27073872
- [Background] Zhu B, Liu JZ, Cauley SF, Rosen BR, Rosen MS. Image reconstruction by domain-transform manifold learning. Nature. 2018 Mar 21;555(7697):487-492. doi: 10.1038/nature25988. PMID 29565357

DOCUMENTS (2):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT05687578/Prot_000.pdf
  • Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT05687578/ICF_001.pdf